CLINICAL TRIAL: NCT03643406
Title: The Influence of Acute Mental Fatigue on Functional Performance Tests of the Lower Limb and Brain Activity in a Healthy Population
Brief Title: The Effect of Mental Fatigue on Lower Limb Functional Performance Tests and Brain Activity in a Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 143201836625
Record Dates: First submitted 2018-08-08; First posted 2018-08-22 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Mental Fatigue; Return to Sport; EEG; Brain Activity; Functional Performance
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Fatigue Condition (Experimental)
  Interventions: Other: Mental Fatigue
- Control Condition (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Mental Fatigue — modified stroop task
  Arms: Mental Fatigue Condition
Other: Control — documentary
  Arms: Control Condition

SUMMARY:
Objective of the study

The main objectives of this project are:

1. To assess the influence of mental fatigue on a return-to-play test battery in healthy population
2. To assess the influence of mental fatigue on brain functioning during a balance and reaction time task in healthy population In a later stage, these experiments could be carried out in a clinical context (e.g. in an ankle sprain population).

The researchers will use a randomized, placebo controlled, counter-balanced, cross-over design.

Thirteen healthy subjects will visit the lab 3 times. On the first visit (familiarisation trial), the investigators will collect the participants' characteristics. The participants will also be familiarized to the procedures and materials of the experiment during this first visit. The second and third visit contain the experimental setup and will proceed as follows: first, the participants will fill in a mental fatigue scale (M-VAS) and motivation scale. Next, the subjects will carry out a functional test battery (hop test, vertical jump test, Y-balance test, and a balance reaction-time test). Session rate of perceived exertion (RPE) is measured to indicate how fatigued the participants feel because of the test battery; also, M-VAS is collected once more. Then, a short cognitive task (Flanker task) is followed by either a long intensive cognitive task (90 minutes Stroop task) or control task (90 minutes documentary). Afterwards, participants have to carry out the Flanker task, fill in M-VAS (2x), perform the same test battery, fill in session RPE and one final fatigue scale (Nasa TLX). Heart frequency and EEG will be measured continuously during the trials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (No neurological/cardiorespiratory/psychological disorders)
* Male and female
* No medication
* Non-smoker
* Between 18 and 35 years old

Exclusion Criteria:

* Back and/or lower extremity injuries during the past 6 months
* Bone/joint abnormalities
* Dizziness, history of loss of consciousness, any inner ear disorders
* Nervous system disorders or dysfunctions
* Uncorrected eye disorders/dysfunctions
* Illness
* Use of medication or any kind of drugs
* Use of alcohol, caffeine and heavy efforts 24 hours before each trial
* Not eating the same meal the night before and the morning of each trial

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Single-leg hop test | Change in single-leg hop test for distance performance: from baseline and 120 minutes after baseline (immediately after the flanker task)
  Single-leg hop test for distance performance
Vertical jump test | Change in vertical jump height performance: from baseline and 120 minutes after baseline (immediately after the flanker task)
  Vertical jump height performance
Y-balance test | Change in Y-balance performance: from baseline and 120 minutes after baseline (immediately after the flanker task)
  Balance and reach performance; participants have to maintain their balance while reaching as far as possible along 3 different directions.
Balance-reaction time test | Change in balance and reaction time performance: from baseline and 120 minutes after baseline (immediately after the flanker task)
  Balance and reaction time performance; participants have to maintain their balance while reacting as fast as possible in 3 different directions.
EEG power spectrum analysis | Change in EEG power spectrum: from baseline and 120 minutes after baseline (immediately after the flanker task)
  Brain activity during the Y-balance test, balance-reaction time test and flanker task will be registered at baseline and immediately after the flanker task

SECONDARY OUTCOMES:
Mental fatigue Visual Analogue Scale (M-VAS) | Change in M-VAS: at baseline, 20 min after baseline (immediately after the first test battery), 120 min after baseline (immediately after the second flanker task) and 135 min after baseline (immediately after the final test battery)
  Subjective measure of mental fatigue (0-10cm; 0 = no mental fatigue; 10 = maximal mental fatigue)
Flanker task | Change in flanker task: at baseline and 90 minutes after baseline (immediately after the mental fatiguing task)
  Objective measure of mental fatigue; reaction time and accuracy give an objective indication of mental fatigue
90-minute stroop task | Change in reaction time and accuracy will be assessed with a 90-min cognitive task; Reaction Time and Accuracy during the 90-min task will be reported as mean reaction time and accuracy during 8 blocks of 11min15sec
  90 minutes mental fatiguing task; reaction time and accuracy give an objective indication of mental fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
individual patient data will not be shared